CLINICAL TRIAL: NCT04127552
Title: Impact of Adrenal IncidenTalomas and Possible Autonomous Cortisol Secretion on Cardiovascular and Metabolic Alterations (ITACA Study)
Brief Title: Impact of Adrenal IncidenTalomas and Possible Autonomous Cortisol Secretion on Cardiovascular and Metabolic Alterations
Acronym: ITACA
Status: Recruiting | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea M. Isidori, Full Professor of Endocrinology, University of Roma La Sapienza
Other Study IDs: ITACA
Record Dates: First submitted 2019-10-06; First posted 2019-10-15 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Adrenal Incidentaloma; Hypercortisolism; Adrenal Tumor
MeSH Terms: conditions — Adrenal incidentaloma; Cushing Syndrome; Adrenal Gland Neoplasms | interventions — Adrenalectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Patients with non-functioning adrenal adenoma: Patients with incidentally discovered adrenal mass with 1mg-DST serum cortisol levels lower than 50 nmol/L
- Patients with pACS receiving conservative management: Patients with incidentally discovered adrenal mass with 1mg-DST serum cortisol levels greater than 50 nmol/L receiving conservative management
- Patients with pACS receiving adrenalectomy: Patients with incidentally discovered adrenal mass with 1mg-DST serum cortisol levels greater than 50 nmol/L receiving adrenalectomy according to the 2016 European Society of Endocrinology guidelines
  Interventions: Procedure: Adrenalectomy
- Healthy controls: Patients without adrenal masses

INTERVENTIONS:
Procedure: Adrenalectomy — Adrenalectomy according to 2016 ESE guidelines
  Groups: Patients with pACS receiving adrenalectomy

SUMMARY:
The investigators hypothesize that cardiovascular and metabolic alterations can occur in patients with adrenal adenomas and possible Autonomous Cortisol Secretion (pACS). Investigators hypothesize that adrenalectomy in selected patients, following the 2016 European Congress of Endocrinology (ECE) guidelines, can improve metabolic parameters and cardiovascular risks and features.

DETAILED DESCRIPTION:
Adrenal incidentalomas are clinically silent masses discovered inadvertently during diagnostic imaging procedures performed for unrelated reasons. Depending on the criteria applied, up to 50% of patients with adrenal incidentalomas may have biochemical evidence of cortisol excess. Possible autonomous cortisol secretion (pACS), as defined in the 2016 European Society of Endocrinology Guidelines, is characterized by a partial, incomplete suppression of the hypothalamic-pituitary-adrenal (HPA) axis without the typical signs of overt cortisol hypersecretion.

Investigators will perform a prospective longitudinal study in patients with adrenal incidentalomas associated with possible autonomous cortisol secretion, aiming to assess the effect of surgical and conservative management on cardiovascular and metabolic features.

Data will be detected at baseline, at 1 and at 5 years follow-up to quantitatively identify the different cardiovascular and metabolic alterations in: (1) patients with non-functioning adrenal adenoma; (2) patients with possible autonomous cortisol secretion receiving conservative management; (3) patients with possible autonomous cortisol secretion receiving adrenalectomy according to the 2016 European Society of Endocrinology guidelines; (4) patients without adrenal masses.

ELIGIBILITY:
Inclusion Criteria:

* Incidentally detected adrenal mass

Exclusion Criteria:

* Patients with overt Cushing's syndrome, pheochromocytoma, Conn syndrome, adrenocortical carcinoma, late-onset congenital adrenal hyperplasia, adrenal metastasis and adrenal hemorrhage
* Patients taking medications influencing glucocorticoid production or metabolism
* Patients with psychiatric diseases or alcohol abuse
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with non-functioning adrenal incidentalomas or adrenal incidentalomas associated with possible autonomous cortisol secretion (subclinical hypercortisolism)
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Echocardiographic Change of Left Ventricular Hypertrophy | at Baseline (T0) and after 1 year (t1) and 5 years (t2)
  Change of Left Ventricular Hypertrophy will be evaluated by transthoracic echocardiography. Patients will be examined in the left lateral decubitus position according to the American Society of Echocardiography guidelines.

SECONDARY OUTCOMES:
Change of arterial stiffness and blood pressure using brachial oscillometric blood pressure waves for a noninvasive estimation. | at Baseline (T0) and after 1 year (t1) and 5 years (t2)
  Perform non-invasive measurement of arterial stiffness
Change of blood pressure using ambulatory blood pressure monitoring blood pressure waves for a noninvasive estimation. | at Baseline (T0) and after 1 year (t1) and 5 years (t2)
  Perform twenty-four-hour systolic and diastolic ambulatory blood pressure monitoring
Change in blood Coagulation Tests | at Baseline (T0) and after 1 year (t1) and 5 years (t2)
  Perform blood sampling for coagulative function
Change in Dual X-Ray Absorptiometry T-score | at Baseline (T0) and after 1 year (t1) and 5 years (t2)
  Bone mineral density change in spine and femur
Radiological evaluation of adrenal mass | at Baseline (T0) and after 1 year (t1) and 5 years (t2)
  Perform adrenal chemical shift MRI or adrenal CT scan (if MRI is contraindicated)
Evaluation of sleep disturbances using questionnaire (PSQI) | at Baseline (T0) and after 1 year (t1) and 5 years (t2)
  Perform the Pittsburgh Sleep Quality Index (PSQI). Sleep disturbances will be evaluated by The Pittsburgh Sleep Quality Index (PSQI). This questionnaire contains 19 self-related questions which are combined to create 7 component scores with a range of 0-3 points (0:no difficulty, 3: severe difficulty). Global score is the result to the addition of all component scores with a range of 0-21 points (0:no difficulty, 21: severe difficulty).
Infectious diseases frequency and severity with modified German Diseases Questionnaire | Baseline (T0), after 1 year (t1) and 5 years (t2)
  Frequencies and severity of infectious diseases will be evaluated by modified Infectious Diseases Questionnaire (GNC).
  This questionnaire includes questions on infectious diseases of upper and lower respiratory tract, gastrointestinal tract, skin and urogenital tract and flu contracted during the previous 12 months. Questions investigate on the number and duration of infections, necessity of antibiotic or antifungal therapy, hospital stay and days of absence from work. Final score represents the frequency of infections.
Quality of life: SF-36-Item Health Survey questionnaire | at Baseline (T0) and after 1 year (t1) and 5 years (t2)
  Quality of life will be evaluated by the Physical Component score and the Mental Component score of the self-administered questionnaire SF-36-Item Health Survey questionnaire.
  This questionnaire measures eight scales: physical functioning, role physical, bodily pain, general health (physical component) and vitality, social functioning, role emotional, mental health (mental component).
  Interpretation of the score will be the following: at each item of the questionnaire corresponds a percentage value (from 0% to 100%). The average of the single items constitutes the scale total percentage (from 0% to 100%); missing data are not considered during calculation. High score defines a more favorable health state.
Psychometric Evaluation: Beck Depression Inventory questionnaire | at Baseline (T0) and after 1 year (t1) and 5 years (t2)
  Psychometric evaluation will be assessed by the score of Beck depression Index: a 21-item measure of depressive symptoms. Each answer is scored on a scale value (from 0 to 3 points). The global score is obtained adding all single scores, with a range of 0-63. Higher score constitutes worse burden of symptoms (0-13: minimal depression, 14-19: mild depression, 20-28: moderate depression, 29-63: severe depression).
Evaluation of sexual dysfunction using FSFI questionnaire in woman | at Baseline (T0) and after 1 year (t1) and 5 years (t2)
  Perform the Female Sexual Function Index (FSFI) questionnaire. This is a 19-item questionnaire that covers six domains: desire, arousal, lubrication, and orgasm, satisfaction, and pain. The ranges of the domain scores are as follows: for desire 1.2 - 6.0, for arousal, lubrication, orgasm and pain 0 - 6.0 and for satisfaction 0.8 - 6.0. The higher scores of the six domains indicate better sexual functioning about that domain. The overall FSFI score is obtained by summing the six domain scores. The overall FSFI scores range from 2.0 to 36.0, with higher scores indicating better sexual functioning.
Evaluation of sexual dysfunction using IIEF questionnaire in man | at Baseline (T0) and after 1 year (t1) and 5 years (t2)
  Perform the International Index of Erectile Function (IIEF) questionnaire in man. The IIEF is an internationally validated test. It is used to assign a score of erectile dysfunction: severe score 1 to 10; moderate score 11 to 16; low to moderate score 17 to 21; Low score 22 to 25; no erectile dysfunction score 26 to 30
Change in insulin resistance calculated with HOMA index | at Baseline (T0) and after 1 year (t1) and 5 years (t2)
  Measurement of HOMA index calculated according to the formula: fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5.
Change in measurement of weight | at Baseline (T0) and after 1 year (t1) and 5 years (t2)
  Measurement of body weight (kg)
Change in blood lipid profile | at Baseline (T0) and after 1 year (t1) and 5 years (t2)
  Measurement of Total Cholesterol, LDL cholesterol, HDL cholesterol, triglycerides

CONTACTS AND LOCATIONS:
Overall Officials: Andrea M Isidori, MD, PHD, Principal Investigator — Sapienza
Locations (1):
- Department of Experimental Medicine, Rome, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Alcubierre D, Ferrari D, Tomaselli A, Moscucci F, Bonaventura I, Francia A, Vozza E, Lospinuso I, Ettorre E, Hasenmajer V, Minnetti M, Sbardella E, Tenuta M, Morelli S, Paganini AM, Isidori AM, Pofi R. Long-Term Cardiac Effects of Adrenalectomy Versus Surveillance in Mild Cortisol Excess: 5-Year Results from the prospective ITACA Study. Eur J Endocrinol. 2026 Jan 23:lvag018. doi: 10.1093/ejendo/lvag018. Online ahead of print. PMID 41572809